CLINICAL TRIAL: NCT00109629
Title: VRC 008: A Phase I Clinical Trial of a Prime-Boost HIV-1 Vaccination Schedule: Multiclade DNA Vaccine, VRC-HIVDNA016-00-VP, Followed by Multiclade Adenoviral Vector Vaccine, VRC-HIVADV014-00-VP, in Uninfected Adult Volunteers
Brief Title: "Prime-Boost" Vaccine Schedule for Prevention of HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050148; 05-I-0148
Record Dates: First submitted 2005-04-29; First posted 2005-05-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-01-22

CONDITIONS: HIV Infections
Keywords: HIV-Negative; Healthy; Immunity; Preventive; Virus; Healthy Volunteer
MeSH Terms: conditions — HIV Infections; Virus Diseases

INTERVENTIONS:
Drug: VRC-HIVDNA016-00-VP
Drug: VRC-HIVADV014-00

SUMMARY:
This study will determine the safety and side effects of two experimental HIV vaccines given in a "prime-boost" schedule. It will also monitor participants for the social impact of being in an HIV vaccine study (e.g., problems with insurance, health care, friends, family, employment, housing, and so forth). The vaccines are VRC-HIVDNA016-00-VP (called the DNA vaccine) and VRC-HIVADV014-00-VP (called the rAd vaccine). The DNA vaccine codes for four HIV proteins. The rAd vaccine is made using an adenovirus (a common virus that causes upper respiratory infections, such as the common cold) that has been modified to contain DNA that codes for three HIV proteins. These vaccines cannot cause HIV or adenoviral infections.

The study will also see if the vaccines cause an immune response; if the injection of the DNA vaccine given using a needle and syringe is similar in safety and immune response to giving them with a needleless injection device called a Biojector 2000; if people who already have antibodies to adenovirus still have an immune response to rAd vaccine; and if there are social harms that result from participating in an HIV vaccine study.

Healthy volunteers between 18 and 50 years of age may be eligible for this 42-week study. Candidates are screened with a medical history, physical examination, blood and urine tests (including pregnancy test for women), and questions regarding sexual behavior and other practices.

Participants receive three injections (shots) of the DNA vaccine and one injection of the rAd vaccine. All injections are given into a muscle in the upper arm (alternating right and left arms with each injection), using a needle and syringe or the needleless Biojector 2000. The first vaccination is given the day of enrollment into the study, and the DNA vaccinations are given about 4 weeks apart from each other, with a minimum of 21 days between injections. The rAd "booster"vaccination is given at Week 24. Participants fill out a diary card at home for 5 days after each vaccination, recording their temperature and any symptoms. They come to the clinic for follow-up 3 days each DNA vaccine injection, and call or return again 7 days after each injection. They call a study nurse 1 or 2 days after the rAd injection.

There are 15 to 18 clinic visits during the course of the study. At each visit, participants are checked for health changes or problems. Blood and urine samples are collected at some visits. Participants are periodically tested for HIV and asked questions about their sexual behavior and drug use and are counseled throughout the study on HIV risk reduction. They are also asked about any social effects they may have experienced as a result of their participation in this study.

DETAILED DESCRIPTION:
Study Design: This is a Phase I randomized study to examine safety and tolerability of, as well as immune response to, a schedule of 3 HIV DNA plasmid vaccinations followed by one HIV adenoviral vector vaccine (rAd) booster. The hypotheses are that: 1) this regimen will be safe for human administration and elicit immune responses to HIV-1; 2) Biojector and Needle/Syringe are both safe to use for IM injection of the DNA vaccine and 3) subjects with both low and high pre-existing adenovirus serotype 5 antibody (Ad5Ab) titer will have a boost in immune response to HIV-1 peptides following the Ad booster vaccination. In this study equal numbers of subjects with high and low Ad5Ab titers will be randomized to receive DNA vaccinations by either needle and syringe (N/S) or by Biojector and then to receive either 1010 PU or 1011 PU rAd booster vaccination in a factorial design. The primary objective is to evaluate the safety and tolerability in humans of the prime-boost vaccination regimen. Secondary objectives are related to evaluation of the immunogenicity of the DNA vaccine when administered by N/S or Biojector, the immunogenicity of the Ad vaccine at two different doses in subjects with high and low pre-enrollment titers of Ad5Ab, the development of adenovirus serotype 5 neutralizing antibody and the social impact of participating in an HIV-1 vaccine trial. Exploratory evaluations of the immunogenicity of the prime-boost regimen are also planned. The preliminary results may serve as the basis for designing studies to provide more definitive answers to questions about method of administration and effect of pre-enrollment Ad5Ab titer on safety of and immune response to the rAd booster vaccination.

Product Description: VRC-HIVDNA016-00-VP is composed of 6 closed, circular DNA plasmids that are each 16.67% (by weight) of the vaccine. Each of the 6 plasmids in this vaccine expresses a single gene product. Plasmids VRC 4401, VRC 4409 and VRC 4404 are designed to express clade B HIV-1 Gag, Pol and Nef, respectively. VRC 5736, VRC 5737, and VRC 5738 are designed to express HIV-1 Env glycoprotein from clade A, clade B, and clade C, respectively. Vaccine vials will be supplied at 4 mg/mL. DNA vaccinations will be 1 mL of vaccine administered intramuscularly using either N/S or the Biojector 2000 Needle-Free Injection Management System. VRC-HIVADV014-00-VP is a recombinant product composed of four non-replicating adenoviral vectors (in a 3:1:1:1 ratio) that code for HIV-1 Gag/Pol polyproteins from clade B and HIV-1 Env glycoproteins from clades A, B, and C. All rAd injections will be administered by N/S.

Subjects: Forty healthy adult volunteers, 18 to 50 years old; 20 subjects with low Ad5Ab (1:500) and 20 subjects with high Ad5Ab (greater than 1:500).

Study Plan: Forty subjects will be randomized in a 1:1 ratio to receive the same vaccination schedule but by two different methods of intramuscular administration (N/S or Biojector), as shown in the schema. The rAd boost will also be randomized to be either 1010 PU or 1011 PU in 1:1 ratio. The rAd boost dosage will be blinded until 6 weeks of safety and immunogenicity evaluations after the rAd boost are completed for all subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

1. 18 to 50 years old.
2. Available for clinical follow-up through Week 42 of the study.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. Complete an Assessment of Understanding prior to enrollment and verbalize understanding of all questions answered incorrectly.
5. Able and willing to complete the informed consent process.
6. Willing to receive HIV test results and willing to abide by NIH guidelines for partner notification of positive HIV results.
7. Willing to donate blood for sample storage to be used for future research.
8. Willing to discuss HIV infection risks and amenable to risk reduction counseling.
9. In good general health without clinically significant medical history.
10. Physical examination and laboratory results without clinically significant findings and a body mass index (BMI) less than 40 within the 28 days prior to enrollment.

    Laboratory Criteria within 28 days prior to enrollment:
11. Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men.
12. White blood cells (WBC) = 3,300-12,000 cells/mm(3).
13. Differential either within institutional normal range or accompanied by site physician approval.
14. Total lymphocyte count greater than or equal to 800 cells/mm(3).
15. Platelets = 125,000 - 550,000/mm(3).
16. Alanine aminotransferase (ALT) less than or equal to 1.25 x upper limit of normal.
17. Serum creatinine less than or equal to upper limit of normal.
18. Normal urinalysis defined as negative glucose, negative or trace protein, and no clinically significant blood in the urine.
19. Negative Food and Drug Administration (FDA)-approved HIV blood test.
20. Negative Hepatitis B surface antigen.
21. Negative anti-HCV (hepatitis C virus antibody) and negative HCV PCR.

    Female-Specific Criteria:
22. Negative beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.
23. A female participant must meet any of the following criteria:

No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

or

Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 42 of the study,

or

Participant agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 42 of the study by one of the following methods:

* condoms, male or female, with or without a spermicide
* diaphragm or cervical cap with spermicide
* intrauterine device
* contraceptive pills or patch, Norplant, Depo-Provera or other FDA-approved contraceptive method
* male partner has previously undergone a vasectomy for which there is documentation.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

Women:

1. Woman who is breast-feeding or planning to become pregnant during the 42 weeks of study participation.

   Volunteer has received any of the following substances:
2. HIV vaccine in a prior clinical trial.
3. Immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis).
4. Blood products within 120 days prior to HIV screening.
5. Immunoglobulin within 60 days prior to HIV screening.
6. Investigational research agents within 30 days prior to initial study vaccine administration.
7. Live attenuated vaccines within 30 days prior to initial study vaccine administration.
8. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration.
9. Current anti-tuberculosis prophylaxis or therapy.

   Volunteer has a history of any of the following clinically significant conditions:
10. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain.
11. Autoimmune disease or immunodeficiency.
12. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.
13. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
14. History of thyroidectomy or thyroid disease that required medication within the past 12 months.
15. Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years.
16. Hypertension that is not well controlled by medication or is more than 145/95 at enrollment.
17. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
18. Syphilis infection that is active or a positive serology due to a syphilis infection treated less than six months ago.
19. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.
20. Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years.
21. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
22. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within five years prior to enrollment, history of a suicide plan or attempt.
23. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.
24. A subject with 3 or more of the 5 health risk factors noted below will be excluded:

    * Current smoker (or quit smoking less than 28 days prior to enrollment)
    * BMI greater than 35
    * Fasting low density lipoprotein (LDL) greater than 159 mg/dL or fasting cholesterol greater than 239 mg/dL
    * Systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg

Fasting blood glucose greater than 125 mg/dL

Note: The fasting blood tests require 8 hours fast prior to the blood draw. The results used for eligibility screening must be from tests completed no more than 12 weeks (84 days) prior to day of enrollment. The individual criteria for BMI (inclusion item 10) and blood pressure (exclusion item 16) must also be met.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2005-04-26; Study Completion 2008-01-22

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Graham BS, Enama ME, Nason MC, Gordon IJ, Peel SA, Ledgerwood JE, Plummer SA, Mascola JR, Bailer RT, Roederer M, Koup RA, Nabel GJ; VRC 008 Study Team. DNA vaccine delivered by a needle-free injection device improves potency of priming for antibody and CD8+ T-cell responses after rAd5 boost in a randomized clinical trial. PLoS One. 2013;8(4):e59340. doi: 10.1371/journal.pone.0059340. Epub 2013 Apr 8. PMID 23577062